CLINICAL TRIAL: NCT03464019
Title: Multi-Centre, Randomized, Double-Blind, Placebo-Controlled, Efficacy, and Safety Study of Etripamil Nasal Spray for the Termination of Spontaneous Episodes of Paroxysmal Supraventricular Tachycardia. NODE 301 and RAPID Studies
Brief Title: Efficacy and Safety of Etripamil for the Termination of Spontaneous Paroxysmal Supraventricular Tachycardia (PSVT).
Acronym: NODE-301
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The closure of the event-driven study was terminated due to the total sample size was reached.
Sponsor: Milestone Pharmaceuticals Inc. (Other)
Collaborators: Medpace, Inc. (Industry); IQVIA Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSP-2017-1138; 2018-000308-41 (EudraCT Number)
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-05

CONDITIONS: Paroxysmal Supraventricular Tachycardia
Keywords: Paroxysmal supraventricular tachycardia; cardiac monitoring; atrioventricular nodal reentrant tachycardia; atrioventricular reciprocating tachycardia; calcium channel blocker administered at home; conversion rate
MeSH Terms: conditions — Tachycardia, Ventricular; Tachycardia, Atrioventricular Nodal Reentry | interventions — etripamil

STUDY DESIGN:
Intervention Model Description: NODE-301 study comprised 6 arms:
  * 2 arms consisting of participants enrolled in Part 1 that treated a perceived episode of PSVT with randomized study drug (etripamil NS 70 mg or placebo) in a 2:1 ratio.
  * 1 arm consisting of participants that only received the Test Dose in Part 1.
  * 2 arms consisting of participants enrolled in Parts 2 and 3 that treated a perceived episode of PSVT with randomized study drug (etripamil NS 70 mg with optional second dose of 70 mg etripamil or placebo) in a 1:1 ratio and could be enrolled in the open-label period to treat an additional PSVT episode with etripamil
  * 1 arm consisting of participants that only received the Test Dose in Parts 2 and 3.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators, and outcomes assessor were blinded to the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: Etripamil 70 mg Single Dose (Experimental): Self-administration of a single dose etripamil 70 mg for a perceived episode of PSVT.
  Interventions: Drug: Etripamil
- Part 1: Placebo Single Dose (Placebo Comparator): Self-administration of a single dose of placebo for a perceived episode of PSVT.
  Interventions: Drug: Placebo
- Part 1: Test dose only (etripamil 70 mg) (Other): Single test dose of etripamil 70 mg in sinus rhythm
  Interventions: Drug: Etripamil Test Dose
- Part 2 & Part 3: Etripamil 70 mg with Optional Second Dose (Experimental): Self-administration of 70 mg etripamil for a perceived episode of PSVT followed 10 minutes later by an optional second dose of 70 mg etripamil, if symptoms persisted. Participants could be enrolled in the open-label period to treat an additional PSVT episode with etripamil.
  Interventions: Drug: Etripamil
- Part 2 & Part 3: Placebo with Optional Second Dose (Placebo Comparator): Self-administration of placebo for a perceived episode of PSVT followed 10 minutes later by an optional second dose of placebo, if symptoms persisted. Participants could be enrolled in the open-label period to treat an additional PSVT episode with etripamil.
  Interventions: Drug: Placebo
- Part 2 & Part 3: Test dose only (etripamil 70 mg + 70 mg) (Other): Repeat Test Dose of etripamil 70 mg (2X 70mg) 10 minutes apart in sinus rhythm
  Interventions: Drug: Etripamil Test Dose

INTERVENTIONS:
Drug: Etripamil — Etripamil administered via the Aptar Pharma Nasal Spray Bidose System, supplied as prefilled devices packaged into child-resistant boxes with instructions for use provided in the study drug box.
  Other Names: MSP-2017
  Arms: Part 1: Etripamil 70 mg Single Dose; Part 2 & Part 3: Etripamil 70 mg with Optional Second Dose
Drug: Placebo — Placebo administered via the Aptar Pharma Nasal Spray Bidose System, supplied as prefilled devices packaged into child-resistant boxes with instructions for use provided in the study drug box.
  Arms: Part 1: Placebo Single Dose; Part 2 & Part 3: Placebo with Optional Second Dose
Drug: Etripamil Test Dose — During the Test Dose, etripamil administered via the Aptar Pharma Nasal Spray Bidose System, supplied as prefilled devices packaged into child-resistant boxes with instructions for use provided in the study drug box.
  Other Names: MSP-2017 Test Dose
  Arms: Part 1: Test dose only (etripamil 70 mg); Part 2 & Part 3: Test dose only (etripamil 70 mg + 70 mg)

SUMMARY:
This was a three-part, multi-center, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of etripamil nasal spray (NS) self-administered by participants who experienced an episode of paroxysmal supraventricular tachycardia (PSVT) in an at-home setting.

NODE-301 Part 1 included participants that received the randomized study drug to treat an episode of PSVT until the 150th positively adjudicated PSVT episode. Part 2 (also referred as the RAPID study) included participants that did not receive the randomized study drug in Part 1 and newly enrolled participants until the 180th positively adjudicated PSVT episode in Part 2. The study continued for approximately 6 months after the 180th positively adjudicated PSVT episode in Part 2 and this extension is referred to as Part 3 (also referred to as RAPID Extension).

DETAILED DESCRIPTION:
NODE-301 was a three-part, multi-center, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of etripamil NS self-administered by participants who experienced an episode of PSVT in an at-home setting. Each episode was documented by an ambulatory Cardiac Monitoring System (CMS) that was placed on the chest by the participants or caregiver when symptoms begin and recorded at least 5 hours of continuous electrocardiogram (ECG).

This was an event-driven study. The study comprised of three parts: Parts 1, 2, and 3.

NODE-301 Part 1 included participants that received the randomized study drug to treat an episode of PSVT until the 150th positively adjudicated PSVT episode (January 15th, 2020). Participants were randomized to etripamil 70 mg or placebo in a 2:1 ratio. Participants had a Test Dose Randomization Visit where they received 70 mg etripamil in sinus rhythm and a Treatment Period during which they could administer the randomized study drug during a perceived episode of PSVT.

Part 2 (also referred as the RAPID study) included participants that did not use the randomized study drug to treat a perceived episode of PSVT before the Part 1 data cutoff and newly enrolled participants. Before randomization in the RAPID study, all participants received a Test Dose of etripamil consisting of an initial dose of etripamil 70 mg followed by a second dose of etripamil 70 mg 10 minutes later to evaluate tolerability and to train participants on the study procedures. After a successful Test Dose, participants in Part 2 were randomized to etripamil or placebo in a 1:1 ratio. When experiencing a PSVT episode, participants were instructed to administer a first dose of randomized study drug (70 mg etripamil or placebo) followed 10 minutes later, if PSVT symptoms persisted, by a second dose of study drug (70 mg etripamil or placebo). After having administered the randomized study drug for a perceived episode of PSVT, participants could enter an open-label period during which they had the possibility to treat a second episode of PSVT with open-label etripamil (70 mg etripamil with optional second dose of 70 mg etripamil).

Part 2 continued until the 180th positively adjudicated PSVT episode (the data on which the primary efficacy analysis of RAPID was conducted) (July 20th 2022). The study continued for approximately 6 months after the 180th positively adjudicated PSVT episode in Part 2 and this extension is referred to as Part 3 (also referred to as RAPID Extension). The design of Parts 2 and 3 were the same and therefore their results are combined in this publication.

NODE-301 study comprised 6 arms:

* 2 arms consisting of participants enrolled in Part 1 that treated a perceived episode of PSVT with randomized study drug (etripamil NS 70 mg or placebo) in a 2:1 ratio.
* 1 arm consisting of participants that only received the Test Dose in Part 1.
* 2 arms consisting of participants enrolled in Parts 2 and 3 that treated a perceived episode of PSVT with randomized study drug (etripamil NS 70 mg with optional second dose of 70 mg etripamil or placebo) in a 1:1 ratio and could be enrolled in the open-label period to treat an additional PSVT episode with etripamil
* 1 arm consisting of participants that only received the Test Dose in Parts 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

Participants who met all of the following criteria were eligible to participate in the study:

1. Male or female participants at least 18 years of age;
2. Electrographically documented history of PSVT (e.g., electrocardiogram [ECG] obtained during an episode of PSVT, Holter monitoring, loop recorder, etc). If participant had a prior ablation for PSVT, participant had to have documented ECG evidence of PSVT post-ablation;
3. History of sustained episodes of PSVT (i.e., typically lasting approximately 20 minutes or longer);
4. Females of childbearing potential who were sexually active with a male partner who were not surgically sterile (i.e., vasectomy) had to agree to use a highly effective form of contraception from the time of signed informed consent until 30 days after the last administration of study drug. Females of childbearing potential had to have a negative serum pregnancy test result at the Screening Visit and at the Final Study Visit, a negative urine pregnancy test at the Test Dose Randomization Visit and had to use a highly effective form of contraception between the visits.

   The following categories defined females who were NOT considered to be of childbearing potential:
   * Premenopausal females with 1 of the following:

     1. Documented hysterectomy,
     2. Documented bilateral salpingectomy or tubal ligation; or
     3. Documented bilateral oophorectomy, or
   * Postmenopausal females, defined as having amenorrhea for at least 12 months without an alternative medical cause;
5. Male participants, except those who were surgically sterile, had to use an approved highly effective form of contraception during the 3 days after any study drug administration; and
6. Signed written informed consent.

Exclusion Criteria:

Participants who met any of the following criteria were excluded from participation in the study:

1. Systolic blood pressure <90 mmHg after a 5-minute rest in sitting position at the Screening Visit or before the Test Dose. In participants treated with a chronic prophylactic drug for PSVT (e.g., beta-blockers, verapamil, and diltiazem), the drug could be stopped for at least the equivalent of 5 half-lives, participants could be rescreened once, and chronic use of the drug could not be restarted after randomization;
2. History of severe symptoms of hypotension, especially syncope, during episodes of PSVT;
3. History of atrial arrhythmia that did not involve the AV node as part of the tachycardia circuit (e.g., atrial fibrillation, atrial flutter, intra-atrial tachycardia);
4. History of allergic reaction to verapamil;
5. Current therapy with digoxin or any Class I or III antiarrhythmic drug, except if these drugs were stopped at least the equivalent of 5 half-lives before the Test Dose Randomization Visit;
6. Current chronic therapy with oral amiodarone, or had taken oral amiodarone within 30 days prior to the Test Dose Randomization Visit;
7. Evidence of ventricular pre-excitation (e.g., delta waves, short PR interval <100 msec, Wolff-Parkinson-White syndrome) on the ECG performed at the Screening Visit or before the Test Dose administration;
8. Evidence of a second- or third-degree AV block on the ECG performed at the Screening Visit or before the Test Dose administration;
9. History or evidence of severe ventricular arrhythmia (e.g., torsades de pointes, ventricular fibrillation, or ventricular tachycardia);
10. Current congestive heart failure defined by the New York Heart Association Class II to IV;
11. History of Acute Coronary Syndrome or stroke within 6 months of screening;
12. Evidence of hepatic dysfunction defined as alanine aminotransferase or aspartate aminotransferase >3 × the upper limit of normal (ULN) or total bilirubin >2 × ULN at the Screening Visit, unless due to Gilbert syndrome;
13. Evidence of End-Stage Renal Disease as determined by an estimated glomerular filtration rate assessed at the Screening Visit of <15 mL/min/1.73m2, or requiring hemodialysis;
14. Females who were pregnant or lactating;
15. Evidence or history of any significant physical or psychiatric condition including drug abuse, which, in the opinion of the Investigator, could jeopardize the safety of participants, or affect their participation in the study. Additionally, the Investigator had the ability to exclude a participant if for any reason the Investigator judged the participant was not a good candidate for the study or would not be able to follow study procedures;
16. Participation in any investigational drug or device study or the use of any investigational drug or device within 30 days of the Screening Visit; or
17. Previously enrolled in a clinical trial for etripamil and received study drug during a perceived episode of PSVT.

Before randomization in the study, all participants received a Test Dose of an etripamil NS dosing regimen (etripamil 70 NS mg in Part 1 and in Parts 2 and 3 an initial dose of etripamil NS 70 mg followed by a second dose of etripamil NS 70 mg not earlier than 10 minutes and not later than 15 minutes after the first dose) to evaluate tolerability and to train participants on the study procedures. Participants who passed the Test Dose were randomized in the NODE-301 (2:1) or RAPID and RAPID Extension (2:1) study. A failure of the Test Dose was considered if participants met any of the following criteria occurring after administration of the either the first or second dose of etripamil NS 70 mg:

1. Any symptoms consistent with clinically severe hypotension such as pre-syncope, medically significant lightheadedness, syncope, nausea, or vomiting;
2. For participants with a pre-Test Dose Systolic Blood Pressure above 100 mmHg:

   1. Decrease in SBP ≥40 mmHg after Test Dose; or
   2. Post-Test Dose SBP <80 mmHg;
3. For participants with a pre-Test Dose SBP between 90 mmHg and 100 mmHg (inclusive):

   a) Post-Test Dose SBP <75 mmHg;
4. Third-degree AV block, Mobitz II second-degree AV block, or Wenckebach with bradycardia ≤40 bpm;
5. New, significant sinus bradycardia Heart Rate ≤40 bpm or sinus pauses (≤3 seconds), if considered by the Investigator to put the participant's safety at risk if either were to occur while not under medical supervision;
6. Any new ventricular arrhythmia considered significant by the Investigator; or
7. Atrial fibrillation, atrial flutter or atrial tachycardia (event lasting longer than 30 seconds);
8. Refusal of second dose of etripamil Test Dose regimen.

Participants who failed the Test Dose proceeded in the study as follows:

* If the Investigator identified a possible reversible cause of the initial Test Dose failure (e.g., concomitant medication such as beta-blocker), a re-challenge with a new Test Dose of etripamil dose regimen was possible after elimination of the reversible cause (e.g., withdrawal of concomitant therapy with the appropriate washout period). Participants could be randomized if they passed the second Test Dose and the cause of the Test Dose failure was eliminated for the duration of the study; or
* If the Investigator could not identify a reversible cause of the initial Test Dose failure, or if the potential cause could not be modified (e.g., necessary antihypertensive drug to control blood pressure), participants could not be randomized and completed a Final Study Visit. Participants who failed the Test Dose are part of the Test Dose Only Population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1097 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bharucha, MD, Study Director — Milestone Pharmaceuticals
Locations (161):
- United States (54):
  - Arizona Arrhythmia Research Center, Phoenix, Arizona
  - Arkansas Cardiology, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Medvin Clinical Research, Cerritos, California
  - North Coast Cardiolog, Encinitas, California
  - Titan Medical Research - Oceanside, Encinitas, California
  - Los Alamitos Cardiovascular, Los Alamitos, California
  - Amicis Research Center - Northridge, Northridge, California
  - RESPIRE Research, Palm Springs, California
  - South Denver Cardiology Associates, P.C, Littleton, Colorado
  - Cardiology Associates of Fairfield County, Norwalk, Connecticut
  - FWD Clinical Research, Boca Raton, Florida
  - Baptist Health Ambulatory Services d/b/a, Jacksonville, Florida
  - United Health Research, LLC, Miami, Florida
  - IACT Health, Columbus, Georgia
  - Piedmont Heart Institute- Fayetteville, Fayetteville, Georgia
  - Piedmont Heart Institute-Fayetteville, Fayetteville, Georgia
  - Georgia Arrythmia Consultants&Research Institute, Macon, Georgia
  - St. Luke's Idaho Cardiology Associates, Boise, Idaho
  - Idaho Catalyst Clinical Research, Idaho Falls, Idaho
  - AMITA Health Medical Group Heart & Vascular Elk Grpve Village, Elk Grove Village, Illinois
  - Parkview Physicians Group - Cardiology, Fort Wayne, Indiana
  - Mercy One Iowa Heart Center, West Des Moines, Iowa
  - Clinical Trials of America, LLC - Monroe, LA, West Monroe, Louisiana
  - MedStar Health Research Institute - Chesapeake Cardiovascular Associates, Baltimore, Maryland
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Revival Research Institute, LLC - Southgate, MI, Southgate, Michigan
  - Mercy Research, St Louis, Missouri
  - Cardiovascular Associates of the Delaware Valley - Elmer, Elmer, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - Atlantic Health System - Morristown Medical Center, Morristown, New Jersey
  - Columbia University, New York, New York
  - New York Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cary Research Group, LLC, Cary, North Carolina
  - Sanger Heart and Vascular Institute, Charlotte, North Carolina
  - The Presbyterian Hospital DBA Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Hatton Institute for Research & Education, Trihealth, Inc. - Cardiology, Cincinnati, Ohio
  - The Ohio State University (OSU) Wexner Medical Center, Columbus, Ohio
  - Rama Research LLC, Marion, Ohio
  - Heart House Research Foundation, LLC, Springfield, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Prisma Health Midlands, Columbia, South Carolina
  - Monument Health Clinical Research, a department of Monument Health Rapid City Hospital, Inc, Rapid City, South Dakota
  - North Texas Research Associates, Allen, Texas
  - Cardiovascular Clinic of North Texas, Denton, Texas
  - Revival Research Institute, LLC, Denton, Texas
  - Apex Trials Group, Fort Worth, Texas
  - Angiocardiac Care of Texas, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Scott & White Memorial Hospital: Baylor Scott & White Research Institute, Temple, Texas
  - Bay Area Heart, Webster, Texas
  - Intermountain Medical Center, Murray, Utah
- Belgium (11):
  - Clinique Du Sud- Luxembourg, Arlon
  - Imelda Hospital, Bonheiden
  - UVC Brugmann University Hospital - Centre Hospitalier Universitaire (CHU), Brussels
  - Universite Libre de Bruxelles (ULB) - Hopital Erasme, Brussels
  - Antwerp University Hospital (UZA), Edegem
  - Grand Hopital de Charleroi (GHdC) - Site Saint-Joseph, Gilly
  - Pharmacy Campus Virga Jesse (losplaats 7), Hasselt
  - University Hospital (UZ) Leuven, Leuven
  - Regional Hospital Centre Citadelle, Liège
  - CHU Ambroise Pare, Mons
  - CHU UCL Namur - Site Godinne, Yvoir
- Canada (20):
  - Libin Cardiovascular Institute of Alberta - University of Calgary, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Medical Arts Health Research Group - North Vancouver, North Vancouver, British Columbia
  - Vancouver Coastal Health Research, Vancouver, British Columbia
  - Victoria Cardiac Arrhythmia Trials, Inc., Victoria, British Columbia
  - University of Manitoba, St Boniface General Hospital, Winnipeg, Manitoba
  - Dalhousie University - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Dawson Road Medical Centre, Guelph, Ontario
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Partners in Advanced Cardiac Evaluation (PACE) Cardiology Clinic, Newmarket, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - The Montreal Heart Institute, Montreal, Quebec
  - CHUM Recherche Cardiologie, Montreal, Quebec
  - McGill University Health Center - Research Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie De Quebec, Québec, Quebec
  - CardioVasc HR, Saint-Jean-sur-Richelieu, Quebec
  - CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec
  - CSSS du Sud de Lanaudiere - Hopital Pierre Le Gardeur, Terrebonne, Quebec
- France (7):
  - CHRU Besancon - Hopital Jean Minjoz, Besançon, Besancon
  - CHU Grenoble-Alpes - Hopital Michallon, La Tronche, Grenoble
  - CHRU de Brest - Hopital de la Cavale Blanche, Brest
  - HCL Hopital Louis Pradel, Bron
  - Hopital Saint-Louis de La Rochelle, La Rochelle
  - CHU de Lille - Institut Cœur Poumon, Lille
  - Centre Hospitalier de Pau, Pau
- Germany (7):
  - Maerkische Gesundheitsholding GmbH - Klinikum Luedenscheid, Lüdenscheid, Ludenscheid
  - Peter Osypka Herzzentrum Munchen, München, Munchen
  - Vivantes Klinikum Neukoelln, Berlin
  - FAZ Dresden-Neustadt GbR, Dresden
  - Kardiologische Praxis, Dresden
  - Kardiologische Gemeinschaftspraxis Papenburg, Papenburg
  - Zentrum fuer Praevention und Rehabilitation, Siegen
- Hungary (7):
  - Dr Lakatos Ferenc Belgyogyaszati-Kardiologiai Maganrendelo, Békéscsaba, Bekescaba
  - Nehezlegzes Ambulancia, Debrecen, Debrecon
  - Del-pesti Centrumkorhaz, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Debreceni Egyetem Klinikai, Debrecen
  - CRU Hungary Kft., Encs
  - Belvarosi Egeszseghaz, Zalaegerszeg
- Netherlands (17):
  - Meander Medisch Centrum - Locatie Amersfoort, Amersfoort
  - Ziekenhuis Rijnstate - Locatie Arnhem, Arnhem
  - Rode Kruis Ziekenhuis, Beverwijk
  - Tergooiziekenhuizen Blaricum, Blaricum
  - Amphia Ziekenhuis - Locatie Breda Molengracht, Breda
  - IJsselland ziekenhuis, Capelle aan den IJssel
  - Reinier de Graaf Gasthuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Slingeland Ziekenhuis, Doetinchem
  - Ziekenhuis Gelderse Vallei, Ede
  - Ropcke-Zweers Ziekenhuis, Hardenberg
  - Treant Zorggroep, Hoogeveen
  - Alrijne Ziekenhuis, Leiderdorp
  - Maastricht University Medical Center, Maastricht
  - Franciscus Gasthuis & Vlietland - Locatie Vlietland, Schiedam
  - Diakonessenhuis - Locatie Utrecht, Utrecht
  - Jeroen Bosch Ziekenhuis, Utrecht
- Poland (15):
  - American Heart of Poland S.A., IV Oddzial Kardiologii Inwazyjnej, Elektrostymulacji i Angiologii, Kędzierzyn-Koźle, Kedzierzyn Kozle
  - Gabinety Daszmed, Krakow, Krakov
  - Kliniczny Szpital Wojewódzki nr 2, Rzeszów, Rzeszów, Rzeszow
  - MICS Centrum Medyczne Torun, Bydgoszcz
  - Centrum Medyczne Kermed, Bydgoszcz
  - Specjalistyczna Praktyka Lekarska, Katowice
  - Prywatny Specjalistyczny Gabinet Internistyczny, Libiąż
  - MEDICOME Sp. z o.o., Oświęcim
  - SP ZOZ Szpital Specjalistyczny w Pulawach, Puławy
  - NZOZ Pro Cordis Sopockie Centrum Badan Kardiologicznych, Sopot
  - Osrodek Badan Klinicznych CLINSANTE S.C., Torun
  - X Oddzial Kardiologii Inwazyjnej, Elektrofizjologii i Elektrostymulacji, Tychy
  - Kardiosystem, Warsaw
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Centralny Szpital Kliniczny, Uniwersytetu Medycznego w Lodzi, Lodz, Łódź Voivodeship
  - Instytut Centrum Zdrowia Matki Polki, Lodz, Łódź Voivodeship
- Spain (23):
  - Martínez Hervás Cardiólogos, Granada, Andalusia
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Hospital Universitario Virgen de la Victoria, Málaga, Malaga
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital General Universitario de Valencia (HGUV), Valencia, Valencia
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Complejo Hospitalario Universitario de Granada - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Universitario Central de Asturias, Oviedo
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitari Sant Joan de Reus, Reus
  - Hospital Universitario la Paz Rua Choupana, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Clínico Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stambler BS, Camm AJ, Alings M, Dorian P, Heidbuchel H, Houtgraaf J, Kowey PR, Merino JL, Mondesert B, Piccini JP, Pokorney SD, Sager PT, Verma A, Wharton JM, Bharucha DB, Plat F, Shardonofsky S, Chen M, Ip JE; RAPID Investigators. Self-administered intranasal etripamil using a symptom-prompted, repeat-dose regimen for atrioventricular-nodal-dependent supraventricular tachycardia (RAPID): a multicentre, randomised trial. Lancet. 2023 Jul 8;402(10396):118-128. doi: 10.1016/S0140-6736(23)00776-6. Epub 2023 Jun 15. PMID 37331368
- [Derived] Stambler BS, Plat F, Sager PT, Shardonofsky S, Wight D, Potvin D, Pandey AS, Ip JE, Coutu B, Mondesert B, Sterns LD, Bennett M, Anderson JL, Damle R, Haberman R, Camm AJ. First Randomized, Multicenter, Placebo-Controlled Study of Self-Administered Intranasal Etripamil for Acute Conversion of Spontaneous Paroxysmal Supraventricular Tachycardia (NODE-301). Circ Arrhythm Electrophysiol. 2022 Dec;15(12):e010915. doi: 10.1161/CIRCEP.122.010915. Epub 2022 Nov 28. PMID 36441560
- [Derived] Stambler BS, Plat F, Sager PT, Lubkov V, Shardonofsky S, Wight D, Chen M, Camm AJ. Rationale for and design of a multicenter, placebo-controlled, phase 3 study to assess efficacy and safety of intranasal etripamil for the conversion of paroxysmal supraventricular tachycardia. Am Heart J. 2022 Nov;253:20-29. doi: 10.1016/j.ahj.2022.06.005. Epub 2022 Jun 18. PMID 35728658

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 431 participants enrolled in Part 1 until the 150th positively adjudicated PSVT episode (15-Jan-2020). After the Part 1 cutoff, 82 participants enrolled in Part 1 transitioned to Part 2 in addition to 624 newly enrolled participants until the 180th positively adjudicated PSVT in Part 2 (20-Jul-2022). The study continued for about 6 months (Part 3) after the Part 2 cutoff with participants waiting for a PSVT episode to arise and 42 newly enrolled participants (27-Feb-2023).
Pre-assignment Details: Participants had to pass a Test Dose before being randomized in the study. 431 participants received the etripamil 70 mg Test Dose before the Part 1 data cutoff. 672 participants received the RAPID etripamil 2x70mg Test Dose before the Part 2 cutoff; including 48 that transitioned from Part 1. An additional 42 participants received the RAPID etripamil 2x70mg Test Dose in Part 3. Participants failing the Test Dose due to safety/tolerability reasons were not randomized in the study.
Groups:
- Placebo: Self-administration of placebo for a perceived episode of PSVT during the randomized treatment period Part 1: single dose. Part 2 and Part 3: single dose followed 10 minutes later by an optional second dose of placebo, if symptoms persisted.
- Etripamil: Self-administration of etripamil for a perceived episode of PSVT during the randomized treatment period.
  Part 1: single dose etripamil 70 mg. Part 2 and Part 3: single dose 70 mg followed 10 minutes later by an optional second dose of etripamil 70 mg, if symptoms persisted.
- Test Dose Only: Single Test Dose of etripamil in sinus rhythm before randomization Part 1: single dose etripamil 70 mg. Part 2 and Part 3: single dose 70 mg followed 10 minutes later by a second dose of etripamil 70 mg.
Period: NODE-301 Part 1
Arm/Group | Placebo | Etripamil | Test Dose Only
Started (Participants received a Test Dose) | 60 | 138 | 233
Participants Randomized | 60 | 138 | 233
Participants in Efficacy Population | 49 | 107 | 0
Completed (Participants in safety population) | 60 | 138 | 0 (Per definition no patient completed the study in the Test Dose only arm as none received the randomized treatment.)
Not Completed | 0 | 0 | 233
Not completed — Withdrawal by Subject | 0 | 0 | 18
Not completed — Ablation | 0 | 0 | 16
Not completed — Test Dose Failure | 0 | 0 | 8
Not completed — Adverse Event | 0 | 0 | 5
Not completed — Physician Decision | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Reason was not provided by the participant | 0 | 0 | 15
Not completed — Transitioned to Part 2 (RAPID) | 0 | 0 | 82
Not completed — Participants did not experienced PSVT before cutoff and did not enroll in Part 2 | 0 | 0 | 80
Period: NODE-301 Part 2 and Part 3
Arm/Group | Placebo | Etripamil | Test Dose Only
Started | 143 (Including participants that transitioned from Part 1-Test Dose Only arm and newly enrolled participants.) | 160 (Including participants that transitioned from Part 1-Test Dose Only arm and newly enrolled participants.) | 445 (Including participants that transitioned from Part 1-Test Dose Only arm and newly enrolled participants.)
Participants Randomized | 143 | 160 | 445
Participants in Efficacy Population | 100 | 114 | 0
Completed (Participants in safety population) | 76 | 81 | 0 (Per definition no patient completed the study in the Test Dose only arm as none received the randomized treatment.)
Not Completed | 67 | 79 | 445
Not completed — Withdrawal by Subject | 5 | 1 | 32
Not completed — Ablation | 8 | 11 | 46
Not completed — Test Dose failure | 0 | 0 | 8
Not completed — Adverse Event | 1 | 3 | 14
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 7
Not completed — Protocol Violation | 0 | 1 | 2
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Prohibited Medication | 1 | 1 | 4
Not completed — Study Terminated by Sponsor | 46 | 61 | 314
Not completed — Reason was not provided by the participant | 5 | 1 | 15

BASELINE CHARACTERISTICS:
Population: Data presented for the overall safety population including participants that received at least one dose of study drug.
Groups:
- Part 1 - Placebo Single Dose: Self-administration of a single dose of placebo for a perceived episode of PSVT during the randomized treatment period.
- Part 1 - Etripamil 70 mg: Self-administration of a single dose of etripamil 70 mg for a perceived episode of PSVT during the randomized treatment period.
- Part 1 - Test Dose Only: Single Test Dose of etripamil 70 mg in sinus rhythm before randomization
- Parts 2 and 3 - Placebo With Optional Second Dose of Placebo: Self-administration of placebo for a perceived episode of PSVT followed 10 minutes later by an optional second dose of placebo, if symptoms persisted, during the randomized treatment period.
- Parts 2 and 3 - Etripamil 70 mg With Optional Second Dose of Etripamil 70 mg: Self-administration of etripamil 70 mg for a perceived episode of PSVT followed 10 minutes later by an optional second dose of etripamil 70 mg, if symptoms persisted, during the randomized treatment period.
- Parts 2 and 3 - Test Dose Only (2X70 mg): Repeat Test Dose of etripamil 70 mg (2X70 mg) 10 minutes apart in sinus rhythm before randomization
- Total: Total of all reporting groups
Arm/Group | Part 1 - Placebo Single Dose | Part 1 - Etripamil 70 mg | Part 1 - Test Dose Only | Parts 2 and 3 - Placebo With Optional Second Dose of Placebo | Parts 2 and 3 - Etripamil 70 mg With Optional Second Dose of Etripamil 70 mg | Parts 2 and 3 - Test Dose Only (2X70 mg) | Total
Number analyzed (Participants) | 60 | 138 | 233 | 143 | 160 | 445 | 1179
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at informed consent signed (years) Population: Participants are included under their respective column.
  years
    Part 1: number analyzed (Participants) | 60 | 138 | 233 | 0 | 0 | 0 | 431
    Part 1 | 55.0 (14.96) | 57.2 (13.58) | 54.1 (15.59) |  |  |  | 55.2 (14.92)
    Parts 2 and 3: number analyzed (Participants) | 0 | 0 | 0 | 143 | 160 | 445 | 748
    Parts 2 and 3 |  |  |  | 55.9 (12.5) | 52.2 (13.9) | 53.9 (14.9) | 53.9 (14.1)
Age, Customized [Mean (Standard Deviation); unit: years] — Population: Participants are included under their respective column.
  years
    Part 1: Age at confirmation of PSVT (years): number analyzed (Participants) | 60 | 138 | 233 | 0 | 0 | 0 | 431
    Part 1: Age at confirmation of PSVT (years) | 53.8 (15.03) | 56.3 (13.69) | 53.2 (15.72) |  |  |  | 54.3 (15.03)
    Parts 2 and 3: Age at confirmation of PSVT (years): number analyzed (Participants) | 0 | 0 | 0 | 143 | 160 | 445 | 748
    Parts 2 and 3: Age at confirmation of PSVT (years) |  |  |  | 54.9 (12.9) | 50.4 (14.5) | 52.5 (14.6) | 52.5 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants are included under their respective column.
  Participants
    Part 1: number analyzed (Participants) | 60 | 138 | 233 | 0 | 0 | 0 | 431
    Part 1: Female | 39 | 92 | 142 |  |  |  | 273
    Part 1: Male | 21 | 46 | 91 |  |  |  | 158
    Parts 2 and 3: number analyzed (Participants) | 0 | 0 | 0 | 143 | 160 | 445 | 748
    Parts 2 and 3: Female |  |  |  | 100 | 112 | 268 | 480
    Parts 2 and 3: Male |  |  |  | 43 | 48 | 177 | 268
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants are included under their respective column.
  Participants
    Part 1: number analyzed (Participants) | 60 | 138 | 233 | 0 | 0 | 0 | 431
    Part 1: Hispanic or Latino | 0 | 5 | 5 |  |  |  | 10
    Part 1: Not Hispanic or Latino | 56 | 129 | 220 |  |  |  | 405
    Part 1: Unknown or Not Reported | 4 | 4 | 8 |  |  |  | 16
    Parts 2 and 3: number analyzed (Participants) | 0 | 0 | 0 | 143 | 160 | 445 | 748
    Parts 2 and 3: Hispanic or Latino |  |  |  | 12 | 11 | 50 | 73
    Parts 2 and 3: Not Hispanic or Latino |  |  |  | 129 | 147 | 384 | 660
    Parts 2 and 3: Unknown or Not Reported |  |  |  | 2 | 2 | 11 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants are included under their respective column.
  Participants
    Part 1: number analyzed (Participants) | 60 | 138 | 233 | 0 | 0 | 0 | 431
    Part 1: American Indian or Alaska Native | 1 | 0 | 0 |  |  |  | 1
    Part 1: Asian | 2 | 5 | 14 |  |  |  | 21
    Part 1: Native Hawaiian or Other Pacific Islander | 0 | 2 | 2 |  |  |  | 4
    Part 1: Black or African American | 4 | 6 | 17 |  |  |  | 27
    Part 1: White | 51 | 120 | 194 |  |  |  | 365
    Part 1: More than one race | 0 | 0 | 0 |  |  |  | 0
    Part 1: Unknown or Not Reported | 2 | 5 | 6 |  |  |  | 13
    Parts 2 and 3: number analyzed (Participants) | 0 | 0 | 0 | 143 | 160 | 445 | 748
    Parts 2 and 3: American Indian or Alaska Native |  |  |  | 0 | 1 | 0 | 1
    Parts 2 and 3: Asian |  |  |  | 5 | 2 | 8 | 15
    Parts 2 and 3: Native Hawaiian or Other Pacific Islander |  |  |  | 0 | 0 | 1 | 1
    Parts 2 and 3: Black or African American |  |  |  | 3 | 5 | 17 | 25
    Parts 2 and 3: White |  |  |  | 131 | 149 | 408 | 688
    Parts 2 and 3: More than one race |  |  |  | 0 | 0 | 0 | 0
    Parts 2 and 3: Unknown or Not Reported |  |  |  | 4 | 3 | 11 | 18
PSVT confirmation duration (years) [Mean (Standard Deviation); unit: years] — Population: Participants are included under their respective column.
  years
    Part 1: number analyzed (Participants) | 60 | 138 | 233 | 0 | 0 | 0 | 431
    Part 1 | 1.7 (4.45) | 1.4 (2.39) | 1.4 (2.39) |  |  |  | 1.4 (2.76)
    Parts 2 and 3: number analyzed (Participants) | 0 | 0 | 0 | 143 | 160 | 445 | 748
    Parts 2 and 3 |  |  |  | 1.6 (3.6) | 2.3 (5.2) | 1.9 (4.2) | 1.9 (4.3)
Number of participant reported PSVT episodes in the past year [Mean (Standard Deviation); unit: episodes] — Population: Information not available for some participants. Participants are included under their respective column.
  episodes
    Part 1: number analyzed (Participants) | 59 | 138 | 232 | 0 | 0 | 0 | 429
    Part 1 | 12.5 (17.91) | 7.8 (7.65) | 6.6 (13.11) |  |  |  | 7.8 (12.60)
    Parts 2 and 3: number analyzed (Participants) | 0 | 0 | 0 | 143 | 160 | 444 | 747
    Parts 2 and 3 |  |  |  | 10.0 (21.1) | 6.8 (15.1) | 5.7 (11.3) | 6.7 (14.5)
Number of participant reported emergency department visits for PSVT in lifetime [Mean (Standard Deviation); unit: emergency department visits] — Population: Information not available for some participants. Participants are included under their respective column.
  emergency department visits
    Part 1: number analyzed (Participants) | 59 | 134 | 230 | 0 | 0 | 0 | 423
    Part 1 | 5.0 (13.17) | 2.7 (3.69) | 2.4 (3.20) |  |  |  | 2.8 (5.87)
    Parts 2 and 3: number analyzed (Participants) | 0 | 0 | 0 | 143 | 160 | 445 | 748
    Parts 2 and 3 |  |  |  | 3.6 (10.3) | 4.3 (14.2) | 2.3 (5.3) | 3.0 (9.0)
Participants with past ablation, n (%) [Count of Participants; unit: Participants] — Population: NODE-301 part 1 did not collect this information.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 143 | 160 | 445 | 748
    Yes |  |  |  | 11 | 13 | 24 | 48
    No |  |  |  | 132 | 147 | 421 | 700
Weight [Mean (Standard Deviation); unit: Kg] — Population: Data not available for some participants. Participants are included under their respective column.
  Kg
    Part 1: number analyzed (Participants) | 60 | 138 | 230 | 0 | 0 | 0 | 428
    Part 1 | 83.99 (20.994) | 82.45 (23.787) | 83.80 (24.149) |  |  |  | 83.39 (23.571)
    Parts 2 and 3: number analyzed (Participants) | 0 | 0 | 0 | 142 | 158 | 430 | 730
    Parts 2 and 3 |  |  |  | 82.7 (19.4) | 81.1 (19.9) | 81.4 (19.3) | 81.6 (19.4)
Height [Mean (Standard Deviation); unit: cm] — Population: Data not available for some participants. Participants are included under their respective column.
  cm
    Part 1: number analyzed (Participants) | 60 | 138 | 230 | 0 | 0 | 0 | 428
    Part 1 | 168.7 (9.12) | 168.8 (10.24) | 169.0 (9.70) |  |  |  | 169.0 (9.6)
    Parts 2 and 3: number analyzed (Participants) | 0 | 0 | 0 | 143 | 159 | 431 | 733
    Parts 2 and 3 |  |  |  | 168.6 (9.4) | 168.7 (9.2) | 169.9 (10.2) | 169.4 (9.9)

OUTCOME MEASURES:

1. Primary Outcome: The Time to Conversion of an Episode of PSVT to Sinus Rhythm (SR) After Study Drug Administration.
Description: The primary efficacy endpoint is defined as an adjudicated termination of a positively adjudicated episode of PSVT (AV nodal reentrant tachycardia or AV reentrant tachycardia determination if possible) and conversion to sinus rhythm (SR) for at least 30 seconds within 5 hours (NODE-301 Part 1), or 30 minutes (NODE-301 Parts 2 and 3) of start of study drug dosing.
Time Frame: NODE-301 Part 1: Within 5 hours of start of study drug dosing. NODE-301 Parts 2 and 3: Within 30 minutes of start of study drug dosing.
Population: In NODE-301 Part 1, the efficacy population consisted of 156 participants (37.2% of the 419 randomized participants).
  In NODE-301 Parts 2 and 3, the efficacy population consisted of 214 participants (29.1% of the 735 randomized participants). The efficacy population was a modified intent-to-treat (mITT) population that included all participants who took study drug to treat an episode of perceived PSVT that was adjudicated by the Independent Adjudication Committee to be confirmed PSVT.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Placebo Single Dose | Part 1 - Etripamil 70 mg | Parts 2 and 3 - Placebo With Optional Second Dose of Placebo | Parts 2 and 3 - Etripamil 70 mg With Optional Second Dose of Etripamil 70 mg
Number analyzed (Participants) | 49 | 107 | 100 | 114
Participants
  Part 1: Participants converted to sinus rhythm within 5 hours: number analyzed (Participants) | 49 | 107 | 0 | 0
  Part 1: Participants converted to sinus rhythm within 5 hours | 36 | 80 |  |
  Part 1: Participants censored: number analyzed (Participants) | 49 | 107 | 0 | 0
  Part 1: Participants censored | 13 | 27 |  |
  Parts 2 and 3: Participants converted to sinus rhythm within 30 minutes: number analyzed (Participants) | 0 | 0 | 100 | 114
  Parts 2 and 3: Participants converted to sinus rhythm within 30 minutes |  |  | 30 | 75
  Parts 2 and 3: Participants censored: number analyzed (Participants) | 0 | 0 | 100 | 114
  Parts 2 and 3: Participants censored |  |  | 70 | 39
Statistical Analysis 1: Comparison: Part 1 - Placebo Single Dose vs Part 1 - Etripamil 70 mg; In Part 1, participants who converted following medical assistance were censored at the time of conversion after medical assistance. Participants who presented missing data from time t to the end were censored at the time of last available data. Participants who did not convert or were not censored before 5 hours were censored at 5 hours; Test type: Superiority; p = 0.1212, Peto-Peto test; Hazard Ratio (HR) = 1.086, 95% CI 2-sided [0.726 to 1.623]
Statistical Analysis 2: Comparison: Parts 2 and 3 - Placebo With Optional Second Dose of Placebo vs Parts 2 and 3 - Etripamil 70 mg With Optional Second Dose of Etripamil 70 mg; In Parts 2 and 3, participants converting after additional medication interventions were censored after the end of the observation period; Test type: Superiority; p < 0.001, Wilcoxon — The threshold for statistical significance was p < 0.05; Hazard Ratio (HR) = 2.857, 95% CI 2-sided [1.868 to 4.371]

ADVERSE EVENTS:
Time Frame: Average of 9.4 months, adverse events were monitored from the time of test dose administration (i.e.,Test Dose Randomization Visit) until study participation was completed (i.e., after the Final Study Visit).
Description: Adverse events were recorded based on the descriptions provided by the participants at every study visit. Adverse events are reported by participants group. For Parts 2 and 3, AEs which occurred after open-label etripamil treatment are included in the columns for placebo and etripamil for completeness.
Groups:
- Parts 2 and 3 - Placebo With Optional Second Dose of Placebo + Open-label Etripamil: Self-administration of placebo for a perceived episode of PSVT followed 10 minutes later by an optional second dose of placebo, if symptoms persisted, during the randomized treatment period. AEs which occur after open-label etripamil treatment are included in this column.
- Parts 2 and 3 - Etripamil 70 mg With Optional Second Dose of Etripamil 70 mg + Open-label Etripamil: Self-administration of etripamil 70 mg for a perceived episode of PSVT followed 10 minutes later by an optional second dose of etripamil 70 mg, if symptoms persisted, during the randomized treatment period. AEs which occur after open-label etripamil treatment are included in this column.
Arm/Group | Part 1 - Placebo Single Dose | Part 1 - Etripamil 70 mg | Part 1 - Test Dose Only | Parts 2 and 3 - Placebo With Optional Second Dose of Placebo + Open-label Etripamil | Parts 2 and 3 - Etripamil 70 mg With Optional Second Dose of Etripamil 70 mg + Open-label Etripamil | Parts 2 and 3 - Test Dose Only (2X70 mg)
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/138 | 0/233 | 0/143 | 0/160 | 1/445
Serious Adverse Events (participants affected / at risk) | 1/60 | 1/138 | 4/233 | 3/143 | 2/160 | 18/445
Other Adverse Events (participants affected / at risk) | 39/60 | 98/138 | 151/233 | 114/143 | 127/160 | 324/445
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - Placebo Single Dose (N=60) | Part 1 - Etripamil 70 mg (N=138) | Part 1 - Test Dose Only (N=233) | Parts 2 and 3 - Placebo With Optional Second Dose of Placebo + Open-label Etripamil (N=143) | Parts 2 and 3 - Etripamil 70 mg With Optional Second Dose of Etripamil 70 mg + Open-label Etripamil (N=160) | Parts 2 and 3 - Test Dose Only (2X70 mg) (N=445)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mesenteric panniculitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Retinal artery occlusion (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - Placebo Single Dose (N=60) | Part 1 - Etripamil 70 mg (N=138) | Part 1 - Test Dose Only (N=233) | Parts 2 and 3 - Placebo With Optional Second Dose of Placebo + Open-label Etripamil (N=143) | Parts 2 and 3 - Etripamil 70 mg With Optional Second Dose of Etripamil 70 mg + Open-label Etripamil (N=160) | Parts 2 and 3 - Test Dose Only (2X70 mg) (N=445)
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 11 | 5 | 8
Atrial fibrillation (Cardiac disorders) | 4 | 0 | 1 | 1 | 2 | 1
Lacrimation increased (Eye disorders) | 9 | 8 | 24 | 28 | 30 | 74
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 6 | 11 | 35
Headache (Nervous system disorders) | 1 | 11 | 11 | 9 | 13 | 38
Dizziness (Nervous system disorders) | 2 | 5 | 13 | 3 | 5 | 23
Dysgeusia (Nervous system disorders) | 3 | 8 | 10 | 5 | 10 | 12
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 15 | 55 | 98 | 58 | 70 | 139
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 24 | 26 | 31 | 42 | 77
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 23 | 29 | 30 | 42 | 59
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 | 23 | 20 | 21 | 31 | 54
Sneezing (Respiratory, thoracic and mediastinal disorders) | 4 | 11 | 10 | 14 | 19 | 38
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 16 | 13 | 14 | 18 | 27
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 9 | 5 | 27
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 4 | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (4):
  • Study Protocol: The RAPID study (NODE-301 Parts 2 and 3) (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT03464019/Prot_000.pdf
  • Study Protocol: NODE-301 Part 1 (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT03464019/Prot_002.pdf
  • Statistical Analysis Plan: The RAPID study (NODE-301 Parts 2 and 3) (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT03464019/SAP_001.pdf
  • Statistical Analysis Plan: NODE-301 Part 1 (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT03464019/SAP_003.pdf